CLINICAL TRIAL: NCT06412406
Title: Comparison Between External Oblique Intercostal Plane Block and the Transversus Abdominis Plane Block in Paraumbilical Hernia Repair as Analgesia for Intraoperative and Postoperative Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Hassan Rashwan, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: paraumbilical hernia
Record Dates: First submitted 2024-02-23; First posted 2024-05-14 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Paraumbilical Hernia
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus abdominis plane (TAP) block (Active Comparator): Group A will include 31 patients to receive TAP block with 20 ml volume on each side (0.25 % bupivacaine)
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- External Oblique intercostal (EOI) block (Active Comparator): Group B will include 31 patients to receive EOI block with 20 ml volume on each side ( 0.25% bupivacaine)
  Interventions: Procedure: External Oblique Intercostal (EOI) block

INTERVENTIONS:
Procedure: External Oblique Intercostal (EOI) block — EOI block technique A linear ultrasound transducer placed in the sagittal plane between the midclavicular and anterior axillary lines at the level of sixth rib, The transducer was then rotated so the cranial end was directed slightly medially and the caudal end laterally to produce a paramedian sagittal oblique view with a short-axis view of the ribs, The following structures were identified, from superficial to deep: subcutaneous tissue, external oblique muscle, intercostal muscles between ribs, pleura, and lung. The skin entry point for the injection was cranial to the sixth rib level just medial to the anterior axillary line, with ultrasound opaque needle advanced in plane from a superomedial-to-inferolateral direction, through the external oblique muscle hydrodissecting the tissue plane between the sixth and seventh ribs, and then the needle was directed caudally toward the eighth rib. and inject 20 ml volume of (0.25 % bupivacaine).
  Arms: External Oblique intercostal (EOI) block
Procedure: Transversus abdominis plane (TAP) block — TAP block technique:
  abdominal skin will be prepared and covered with sterile drapes. The needle can be introduced by multiple punctures along the oblique subcostal line from the xiphoid process towards the anterior part of the iliac crest (18) . Thus, LA will be injected in the TAP along this line provides both upper and lower abdominal wall analgesia. The OSCTAP block more consistently covers L1 dermatome. After negative aspiration, a test injection with 1 ml of 0.9% normal saline will be performed to confirm the needle location. and ingect 20 ml volume of (0.25 % bupivacaine). If the intended sensation will not decreased in surgical dermatomes after 30 min, the patient will be regarded to have a failed block and will be excluded from the study.
  Arms: Transversus abdominis plane (TAP) block

SUMMARY:
AIM OF STUDY:

Comparison between effect of external oblique intercostal plane block and the Oblique subcostal transversus abdominis plane block in paraumbilical hernia repair as analgesia for intraoperative and postoperative pain.

DETAILED DESCRIPTION:
A paraumbilical hernia is a hole in the connective tissue of the abdominal wall in the midline with close approximation to the umbilicus. If the hole is large enough there can be protrusion of the abdominal contents, including omental fat and/or bowel. These defects are usually congenital and are not noticed until they slowly enlarge over an individual's life time and abdominal contents herniate through the hole creating either pain or a visible lump on the abdominal wall. If abdominal contents get incarcerated (or stuck) in the hole this can cause pain. If the abdominal contents become strangulated by losing their blood supply from pinching or twisting those tissue will die. If it is omental fat this will cause pain and could potentially lead to an infection. If the strangulated contents are bowel then in addition to pain the individual will develop a bowel obstruction. And if the dead bowel is not surgically removed in an emergent fashion the condition could be fatal.

Postoperative pain is the major obstacle for early postoperative ambulation and increases the risk of venous thromboembolism and respiratory complications and prolongs the hospital stay. This pain is routinely managed using opiates, which are associated with several side effects, including excessive sedation and postoperative nausea and vomiting (PONV) which may increase hospital stay durations. Transversus abdominis plane (TAP) block is a regional anesthetic technique that has gradually become an alternative for postoperative pain control during laparoscopic abdominal surgeries. It involves the infusion of local anesthetic into the fascial plane of the abdominal wall.

the subcostal transversus abdominis plane block (TAP) targets the upper abdominal wall.

The EOI block represents an important modification that cover the upper lateral abdominal wall.

Oblique subcostal transversus abdominis plane (OSCTAP) block is an US-guided regional anesthesia technique that anesthetizes the nerves of the lower and upper anterior abdominal wall,specifically from T6 to L1. The OSCTAP has been described that can be performed to provide analgesia for abdominal surgery extending above the umbilicus.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years with a body mass index (BMI) of 18-35 kg/m2
2. patients with the American Society of Anesthesiologists (ASA) physical status I/II
3. Patients scheduled for elective paraumbilical hernia

Exclusion Criteria:

* 1-Known hypersensitivity to the study drugs. 2-Body Mass Index > 40 kg/m2. 3- Inability to accurately describe postoperative pain to investigators. 4-Opioid tolerance or dependence. 5-Preexisting history of chronic pain. 6-History of renal, liver, cardiac, neuropsychiatric disorder problems. 7-Bleeding or coagulation abnormality. 8-Patients who received any analgesic 24 h before surgery 9-Patients who have difficulty understanding the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
The effect between external oblique intercostal plane block and the transversus abdominis plane block in paraumbilical hernia repair as analgesia for intraoperative and postoperative pain according to numeric rating score (NRS) | baseline
  numeric rating scale : from 0 to 10 0 : no pain
  1 - 3 : mild pain 4 - 6 : moderate pain 7 - 9 : severe pain 10 : worst pain possible

SECONDARY OUTCOMES:
time of the first opioid request | baseline
  time of the first opioid request all over 24 hours postoperatively.
Heart rate | baseline
  heart rate will be recorded at time 0 then every 15 minutes in the first 2 hours, then at 6, 12, 24 hours postoperatively.
Mean arterial blood pressure | baseline
  mean arterial blood pressure will be recorded at time 0 then every 15 minutes in the first 2 hours, then at 6, 12, 24 hours postoperatively.
time to start ambulation | baseline
  time of the patient first movement will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nawal A Gadelrab, Professor, Study Chair — Assiut University; Abdelrahim M Mohamed, Professor, Study Chair — Assiut University; Mohamed G Hassan, Resident, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Elsharkawy H, Maniker R, Bolash R, Kalasbail P, Drake RL, Elkassabany N. Rhomboid Intercostal and Subserratus Plane Block: A Cadaveric and Clinical Evaluation. Reg Anesth Pain Med. 2018 Oct;43(7):745-751. doi: 10.1097/AAP.0000000000000824. PMID 30169476
- [Background] Desai N, El-Boghdadly K, Albrecht E. Epidural vs. transversus abdominis plane block for abdominal surgery - a systematic review, meta-analysis and trial sequential analysis. Anaesthesia. 2021 Jan;76(1):101-117. doi: 10.1111/anae.15068. Epub 2020 May 8. PMID 32385856
- [Background] Qin C, Liu Y, Xiong J, Wang X, Dong Q, Su T, Liu J. The analgesic efficacy compared ultrasound-guided continuous transverse abdominis plane block with epidural analgesia following abdominal surgery: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Feb 28;20(1):52. doi: 10.1186/s12871-020-00969-0. PMID 32111162
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Gan TJ, Diemunsch P, Habib AS, Kovac A, Kranke P, Meyer TA, Watcha M, Chung F, Angus S, Apfel CC, Bergese SD, Candiotti KA, Chan MT, Davis PJ, Hooper VD, Lagoo-Deenadayalan S, Myles P, Nezat G, Philip BK, Tramer MR; Society for Ambulatory Anesthesia. Consensus guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2014 Jan;118(1):85-113. doi: 10.1213/ANE.0000000000000002. PMID 24356162
- [Background] Elsharkawy H, Pawa A, Mariano ER. Interfascial Plane Blocks: Back to Basics. Reg Anesth Pain Med. 2018 May;43(4):341-346. doi: 10.1097/AAP.0000000000000750. PMID 29561295
- [Background] Sondekoppam RV, Brookes J, Morris L, Johnson M, Ganapathy S. Injectate spread following ultrasound-guided lateral to medial approach for dual transversus abdominis plane blocks. Acta Anaesthesiol Scand. 2015 Mar;59(3):369-76. doi: 10.1111/aas.12459. Epub 2015 Jan 13. PMID 25582299
- [Background] Borglum J, Jensen K, Christensen AF, Hoegberg LC, Johansen SS, Lonnqvist PA, Jansen T. Distribution patterns, dermatomal anesthesia, and ropivacaine serum concentrations after bilateral dual transversus abdominis plane block. Reg Anesth Pain Med. 2012 May-Jun;37(3):294-301. doi: 10.1097/AAP.0b013e31824c20a9. PMID 22476239
- [Background] Tulgar S, Senturk O, Selvi O, Balaban O, Ahiskalioglu A, Thomas DT, Ozer Z. Perichondral approach for blockage of thoracoabdominal nerves: Anatomical basis and clinical experience in three cases. J Clin Anesth. 2019 May;54:8-10. doi: 10.1016/j.jclinane.2018.10.015. Epub 2018 Oct 31. No abstract available. PMID 30388604
- [Background] Hutchins J, Delaney D, Vogel RI, Ghebre RG, Downs LS Jr, Carson L, Mullany S, Teoh D, Geller MA. Ultrasound guided subcostal transversus abdominis plane (TAP) infiltration with liposomal bupivacaine for patients undergoing robotic assisted hysterectomy: A prospective randomized controlled study. Gynecol Oncol. 2015 Sep;138(3):609-13. doi: 10.1016/j.ygyno.2015.06.008. Epub 2015 Jun 6. PMID 26056753
- [Background] Hebbard PD, Barrington MJ, Vasey C. Ultrasound-guided continuous oblique subcostal transversus abdominis plane blockade: description of anatomy and clinical technique. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):436-41. doi: 10.1097/aap.0b013e3181e66702. PMID 20830871
- [Background] Cosarcan SK, Ercelen O. The analgesic contribution of external oblique intercostal block: Case reports of 3 different surgeries and 3 spectacular effects. Medicine (Baltimore). 2022 Sep 9;101(36):e30435. doi: 10.1097/MD.0000000000030435. PMID 36086688
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Marhofer P, Harrop-Griffiths W, Kettner SC, Kirchmair L. Fifteen years of ultrasound guidance in regional anaesthesia: part 1. Br J Anaesth. 2010 May;104(5):538-46. doi: 10.1093/bja/aeq069. Epub 2010 Apr 2. PMID 20364022
- [Background] Soliz JM, Lipski I, Hancher-Hodges S, Speer BB, Popat K. Subcostal Transverse Abdominis Plane Block for Acute Pain Management: A Review. Anesth Pain Med. 2017 Oct 20;7(5):e12923. doi: 10.5812/aapm.12923. eCollection 2017 Oct. PMID 29696110